CLINICAL TRIAL: NCT05442541
Title: Üreme çağındaki kadınlarda menstrüel Iyilik Halinin değerlendirilmesi Saha Anket çalışması/Evaluation of Menstrual Well-being in Women of Reproductive Age, Field Survey Study
Brief Title: Menstrual Wellbeing in Woman Living in Turkey; an Epidemiological Study
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Collaborators: Turkish Endometriosis and Adenomyosis Society (Unknown); IPSOS (Industry)
Responsible Party: Principal Investigator, Elif Cansu Gundogdu, Principal Investigator, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: 2021/514/216/15
Record Dates: First submitted 2022-01-12; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Menstrual Problem; Quality of Life
Keywords: menstrual wellbeing; reproductive age; oral contraceptive; endometriosis
MeSH Terms: conditions — Menstruation Disturbances; Endometriosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: not included any interventions(Evaluation of menstrual well-being in women of reproductive age, field survey study) — This is a prospective cross-sectional analytical study conducted through a questionnaire.

SUMMARY:
Women with endometriosis in our country and around the world face various difficulties during their menstrual periods in reproductive age. While some of these difficulties are caused by the environment, some of them are due to the insufficient development of personal consciousness. In our study, we aim to reveal the perspective of individuals and society on the menstrual period. Our primary aim in our study is to understand what kind of problems are experienced in different regions of our country during the menstrual period for women and how they are spent. Secondly, the effect of this period on women's quality of life will be examined.

DETAILED DESCRIPTION:
Our research will be conducted between January 1, 2022, and February 1, 2022, in 7 different regions of our country, by asking questions to women of reproductive age from different groups. Each participant will be asked to answer the survey questions and the results will be analyzed. The survey will be done face to face. The questionnaire contains questions about women's socio-demographic data, their perspectives on their menstrual period, their information about endometriosis, and their perspectives on pads and birth control pills. Menstruating women of reproductive age between the ages of 18- 45 will be included in this study. As a result of the study, the problems experienced by women of reproductive age in different regions will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Menstruating women of reproductive age between the ages of 18- 45 will be included in this study.

Exclusion Criteria:

* Women with a history of hematological disease, cardiovascular disease, malignancy, advanced renal failure, active infection, diabetes mellitus, and pregnant women will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Menstruating women of reproductive age between the ages of 18- 45 will be included in this study
Study Population: Menstruating women of reproductive age between the ages of 18- 45 will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1829 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Disparities in menstrual hygiene and well-being between 7 regions of Turkey in women of reproductive age with a questionnaire | 1 month
  In this study, the effect of the menstrual period on the quality of life of 1829 women living in seven different geographical regions of our country will be examined through a questionnaire. The goal of this study is to evaluate the menstrual well-being of women living in different regions of our country.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Kale, Prof.Dr., Study Director — Kartal Dr. Lutfi Kirdar Research and Training Hospital
Locations (1):
- Kartal Dr. Lutfi Kirdar Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet.